CLINICAL TRIAL: NCT00004557
Title: Models of Disordered Knowledge and Memory Systems in Dementia and Related Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 920075; 92-M-0075
Record Dates: First submitted 2000-02-08; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-02

CONDITIONS: Dementia
Keywords: Attention; Cognition; Dementia; Memory; Object Recognition; Spatial Processes
MeSH Terms: conditions — Dementia

SUMMARY:
Patients with Alzheimer's disease (AD) perform poorly on tasks dependent on access to, and utilization of, previously acquired knowledge and skills. It has been commonly assumed that impaired knowledge in AD, as well as in other patients with cortical lesions, is due to an actual loss or disorganization of a specific knowledge base or system. This hypothesis has, however, recently been called into question by data from tasks that purport to tap knowledge on a more automatic and implicit level. For example, although AD patients are impaired on object naming and verbal fluency tasks, they show a normal pattern of semantic facilitation on reaction time based priming tasks. In fact, the level of facilitation or activation on these tasks has often been reported to be greater in AD patients than in normal individuals. These and similar data have been used to support arguments that performance decrements in AD patients are due to deficits in attentional and/or retrieval processes rather than a degradation of knowledge stores. The central focus of this project will be to test a model of the semantic representations of object that predicts increased facilitation or hyperpriming in AD patients as a result of degraded representations. The relationship between performance on on-line priming tasks, visual attention and spatial processes, and explicit and implicit measures of memory also will be examined. In addition to normal controls, patients with cognitive and memory impairments, but without semantically-based naming difficulties (elderly depressed, Huntington's disease, Korsakoff's disease) will serve as controls for overall slowness of response and degree of explicit memory deficit.

DETAILED DESCRIPTION:
Patients with Alzheimer's disease (AD) perform poorly on tasks dependent on access to, and utilization of, previously acquired knowledge and skills. It has been commonly assumed that impaired knowledge in AD, as well as in other patients with cortical lesions, is due to an actual loss or disorganization of a specific knowledge base or system. This hypothesis has, however, recently been called into question by data from tasks that purport to tap knowledge on a more automatic and implicit level. For example, although AD patients are impaired on object naming and verbal fluency tasks, they show a normal pattern of semantic facilitation on reaction time based priming tasks. In fact, the level of facilitation or activation on these tasks has often been reported to be greater in AD patients than in normal individuals. These and similar data have been used to support arguments that performance decrements in AD patients are due to deficits in attentional and/or retrieval processes rather than a degradation of knowledge stores. The central focus of this project will be to test a model of the semantic representations of object that predicts increased facilitation or hyperpriming in AD patients as a result of degraded representations. The relationship between performance on on-line priming tasks, visual attention and spatial processes, and explicit and implicit measures of memory also will be examined. In addition to normal controls, patients with cognitive and memory impairments, but without semantically-based naming difficulties (elderly depressed, Huntington's disease, Korsakoff's disease) will serve as controls for overall slowness of response and degree of explicit memory deficit.

ELIGIBILITY:
Subjects will include:

Patients assigned a diagnosis of probable Alzheimer's disease meeting NINCDS-ADRDA and DSM-III-R criteria.

Patients with other neuropsychiatric illness (i.e., depression, Korsakoff's disease, Huntington's disease).

Normal controls.

Subjects must not have major concomitant illness.

All patients will be drug-free for at least 2 weeks whenever possible. Concurrent use of some medications (i.e., diuretics or antibiotics) will be allowed only after careful review by the investigators.

Normal control subjects will be without a history of or present psychiatric or neurological illness.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 650
Dates: Start 1992-01; Study Completion 2000-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Balota DA, Duchek JM. Semantic priming effects, lexical repetition effects, and contextual disambiguation effects in healthy aged individuals and individuals with senile dementia of the Alzheimer type. Brain Lang. 1991 Feb;40(2):181-201. doi: 10.1016/0093-934x(91)90124-j. PMID 2036582
- [Background] Bayles KA, Tomoeda CK. Confrontation naming impairment in dementia. Brain Lang. 1983 May;19(1):98-114. doi: 10.1016/0093-934x(83)90057-3. PMID 6222782
- [Background] Butters N, Granholm E, Salmon DP, Grant I, Wolfe J. Episodic and semantic memory: a comparison of amnesic and demented patients. J Clin Exp Neuropsychol. 1987 Oct;9(5):479-97. doi: 10.1080/01688638708410764. PMID 2959682